CLINICAL TRIAL: NCT04866836
Title: A Single-arm, Open, Exploratory Clinical Study of Tislelizumab Combined With Radiotherapy as the Second-line Treatment of Advanced Biliary Malignant Tumors
Brief Title: A Study of Tislelizumab Combined With Radiotherapy as the Second-line Treatment of Advanced Biliary Malignant Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated due to difficulties in recruitment.
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hepatobiliary Center
Record Dates: First submitted 2021-04-16; First posted 2021-04-30 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiotherapy; spartalizumab

STUDY DESIGN:
Intervention Model Description: To observe and evaluate the effectiveness and safety of tislelizumab combined with radiotherapy in the treatment of patients with advanced biliary malignancies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab combined with radiotherapy (Experimental): To observe and evaluate the effectiveness and safety of tislelizumab combined with radiotherapy in the treatment of patients with advanced biliary malignancies.
  Interventions: Combination Product: Radiotherapy

INTERVENTIONS:
Combination Product: Radiotherapy — Patients who meet the criteria for enrollment first receive radiotherapy, either IMRT or SBRT, and the relative biological effect dose is> 40Gy. On the 7th day (±3 days) after radiotherapy, start to give tislelizumab 200 mg, IVD, q3w, and continue the treatment until disease progression, unacceptable toxic radiotherapy, death or meet the description in the protocol Any discontinuation criteria shall be subject to whichever occurs firs
  Other Names: PD-1 monoclonal antibody

SUMMARY:
Biliary tract cancer (BTC) accounts for 4% of the malignant tumors of the digestive system, and the incidence has increased significantly in recent years. For advanced malignant tumors of the biliary tract, the existing treatment methods are very limited and the effective rate is low. At present, gemcitabine combined with platinum therapy is the first-line standard treatment for advanced biliary tract cancer. In recent years, tumor immunotherapy has made huge breakthroughs. There are also research attempts in advanced biliary tract cancer. A study published in the international top medical journal NEJM in 2015 showed that PD-1 monoclonal antibody treatment has mismatch gene repair defects. Patients with advanced biliary tract tumors have a higher curative effect. It suggests that PD-1 monoclonal antibody is worthy of in-depth study in the treatment of biliary tract tumors.

In the previous clinical studies of PD-1 in the treatment of biliary tract tumors conducted by our center, it was observed that the tumor control of some patients was stable with the combination of immunotherapy and radiotherapy. In view of the observations in the clinical research of our unit, relevant case reports, and the mechanism of the combination of radiotherapy and immunotherapy, we speculate that in patients with biliary tract cancer, radiotherapy and immunotherapy have a certain combined sensitization effect. Therefore, it is planned to carry out clinical research on the second-line treatment of advanced biliary tract cancer with radiotherapy and immunotherapy.

This study will explore the effectiveness and safety of tislelizumab combined with radiotherapy in the treatment of patients with advanced biliary malignant tumors (BTC) in second-line and above, with a view to improving the therapeutic effect of biliary tract tumors.

DETAILED DESCRIPTION:
Patient recruitment Research and discussion by the MDT team of the Department of Hepatobiliary Surgery of our center: Choose pathologically confirmed malignant tumors of the biliary tract that are inoperable or recurring after surgery, including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer; patients with non-extensive metastases, after full communication with the patient, The patients joined the study after signing the informed consent form voluntarily.

During the study Each period of the test period is defined as 3 weeks. After starting tislelizumab, tumor imaging evaluation will be performed every 6 weeks (±7 days). Until the disease progresses or treatment ends.

Radiation Therapy We use intensity-modulated radiotherapy (IMRT) or stereotactic radiotherapy (SBRT) based on comprehensive factors such as the location of the lesion, the irradiation volume, the volume of the normal liver, liver function, and the general condition of the patient. The divided dose is within 3-7.5Gy. The number of divisions is between 2-15. Daily irradiation from Monday to Friday/week, or every other day on Monday, Wednesday, and Friday/week, strive to achieve a relative biological dose (BED) of more than 40Gy, and the exposure to organs at risk within the accepted range.

medical treatment On the 7th day (±3 days) after the start of radiotherapy, tislelizumab was given 200 mg, IVD, q3w, and continued treatment until disease progression, unacceptable toxic radiotherapy, death or meet any discontinuation criteria described in the protocol.

Follow up Safety follow-up Regardless of whether the patient starts a new anti-tumor therapy, the patient should be contacted 30 days (± 7 days) after the last dose of tislelizumab to assess irAE and concomitant medications.

Survival follow-up After the study treatment is terminated, the survival status of all patients and more information on anti-cancer treatment will be followed up, patient medical records and/or outpatient visits. After the treatment ends, the visit will be conducted approximately once every 1 month (±7 days) until the patient died, was lost to follow-up, withdrawn informed consent, or the sponsor completed the study. The situation of each survival follow-up should be recorded in the follow-up form in detail.

Effectiveness evaluation Tumor imaging examinations will be performed 28 days before the first administration of the study drug. During the study period, tumor imaging examinations were performed every 6 weeks (±7 days) during the treatment cycle of tislelizumab.The screening evaluation and each follow-up evaluation must include contrast-enhanced computed tomography (CT) or contrast-enhanced magnetic resonance imaging (MRI) of the chest, abdomen, and pelvis. Other known or suspected lesions must be included in the imaging evaluation. Assessment of the lesions using the same contrast agent program, but in special circumstances, if MRI is selected as the tumor assessment for the entire study process, in the chest imaging assessment, chest non-thoracic imaging should be performed. All known lesions must be recorded at the time of screening, and the assessment must be repeated for each subsequent tumor assessment.

After the first remission (CR or PR), tumor remission should be confirmed ≥ 4 weeks after the first remission or at the next planned evaluation time point.

Safety assessment Adverse events (AE) and Serious adverse event (SAE) AE is defined as any adverse physical signs (including abnormal laboratory test results), symptoms or diseases (new or worsening) that are related to the study treatment in time, regardless of whether it is considered to be related to the study drug.

If an AE or SAE occurs, the investigator is responsible for reviewing all records related to the AE or SAE (such as hospital history records, laboratory test results, and diagnostic reports). The investigator will then record all information related to the AE or SAE in the case report form (CRF).

Disease progression Disease progression is defined as the deterioration of the subject's condition caused by the primary tumor targeted by the experimental drug.The appearance of new metastases relative to the original tumor or the progression of the original metastases are considered to be disease progression. Events that are life-threatening due to symptoms and signs of disease progression, require hospitalization or prolong hospitalization, or cause permanent or severe disability/dysfunction/affect work ability, and congenital abnormalities or birth defects are not reported as SAEs for accelerated reporting. Death due to symptoms and signs of disease progression is reported as an accelerated SAE.

SAE should record in detail the symptoms, severity, correlation with the test drug, time of occurrence, treatment time, measures taken, time and method of follow-up, and outcome. If the intensity of an ongoing SAE or its relationship with the test drug changes, a follow-up report should be submitted immediately.

Data collection and data management This study will use the case report form (CRF) to collect and manage research data.

Data collection This research uses CRF table to collect research data. Researchers and CRC collect relevant data in detail. The clinical research quality control personnel conduct corresponding quality control.

Data management and quality control In order to ensure the authenticity and reliability of clinical trial data and improve the quality of clinical data, clinical monitors will follow standard operating procedures to review the completeness, consistency and accuracy of the trial data in the clinical database and provide guidance during the trial project. The personnel of the research institution shall make necessary supplements or corrections to the problem data. Clinical monitors or data managers will question the questionable data to PI or CRC in the form of an electronic questioning form. PI or CRC must respond to the questioning and make corrections or explanations to the questioned data. The person in charge of medicine and data management personnel conduct regular consistency comparisons of SAE.

At the end of the test project, data management personnel and medical personnel will perform final quality control on all data in the database, summarize all program deviations and program violations that occurred during the test, and hold a data verification meeting. After the data in the database meets the quality requirements, the database will be locked and tested, and the data management staff will export the data for data analysis by the statistics department.

Data review and monitoring of research institutions Researchers must keep the original documents of each patient participating in the trial, including research medical records and visit records. The researcher must confirm that all relevant original documents can be monitored to verify that they are consistent with the CRF content.

Data analysis and statistical methods The detailed summary and statistical analysis methods for the data collected by this research will be included in the statistical analysis plan (SAP), which will be finalized and filed by the sponsor. Any changes to this research plan, if determined by the sponsor or the main investigator, have a significant impact on the statistical analysis plan, SAP needs to be revised to be consistent with the research plan.

Determination of sample size This study is an exploratory clinical study. It is expected that 20 patients will be enrolled. If objective remission of 5 or more cases can be obtained, the combined treatment method is considered to have the effect of increasing sensitivity, and follow-up clinical studies are recommended.

Analyze the population Full Analysis Set (FAS): An analysis set determined in accordance with the principle of intentional analysis. All subjects who are enrolled and have at least one treatment record will be included in this analysis set. The full analysis set is the main effectiveness analysis set.

In line with the plan set (PPS): a subset of the full analysis set. Subjects who have violated the protocol and judged that the violation has a significant impact on the efficacy will be excluded from this set.

Definition of the evaluable population: All subjects who meet the following criteria have received at least one treatment with tislelizumab and have received one tumor evaluation. If the curative effect reaches CR or PR, the subject must confirm the curative effect.

Safety analysis set (SS): All subjects who have been enrolled and have at least one treatment record will be included in the safety analysis set.

Exploratory index analysis set: All subjects who are included in the group and who have used the trial drug at least once and obtained tumor biopsy samples will be included in this analysis set.

Statistical analysis General analysis Unless otherwise specified, continuous variables in this study are summarized by mean, standard deviation, median, maximum, and minimum; categorical variables are summarized by frequency and percentage; time-event data are estimated by Kaplan-Meier method Survival rate and median survival time.

Effectiveness analysis Tumor evaluation will be made by investigators based on RECIST v1.1. The evaluation data will be based on the following response indicators: complete remission (CR), partial remission (PR), stable disease (SD), disease progression (PD) and non-evaluable (NE). The survival distribution of OS will be estimated based on the Kaplan-Meier (KM) method, and the median OS and a bilateral 95% confidence interval will be calculated. In addition, the KM method is used to estimate the survival probability at different time nodes (6/9/12 months), and the corresponding 95% confidence interval is calculated.

The survival distribution of progression-free survival (PFS) will be estimated based on the Kaplan-Meier (KM) method, and the median PFS and the two-sided 95% confidence interval will be calculated.

The objective response rate (ORR) and disease control rate (DCR) will use the Clopper-Pearson method to calculate the 95% confidence interval for the percentage of cases.

Security Analysis The analysis of AEs will be based on the safety analysis set. Data analysis will include, but not limited to, grouping and calculating the incidence of adverse reactions; the sub-system will list the frequency and frequency of adverse reactions, the calculation percentage, and a detailed list of various AE cases. The analysis will be stated in the statistical analysis plan.

Case shedding All subjects who have filled out the informed consent form and screened qualified to enter the trial have the right to withdraw from the clinical trial at any time. Regardless of when and for any reason, as long as the subjects who have not completed one cycle of the clinical trial and cannot be evaluated for safety and effectiveness, they are all dropped cases (after being enrolled in the group due to disease progression and clear medical evidence, they will not be regarded as dropped out. ). When the subject falls off, the researcher must fill in the reason for the fall off in the CRF, complete the assessment items that can be completed, and carefully fill in the last visit record in the CRF. Those who fall off due to adverse reactions and are determined to be related to the test drug after follow-up should be recorded in the CRF and the investigator should be notified. If the subject has completed a complete cycle and has a detailed record, statistical analysis should be made during the safety evaluation.Subjects who withdraw from the study cannot re-enter the study, and their number cannot be used again.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of Advanced biliary malignancy
* The expected survival period is ≥3 months
* Patients with non-extensive metastases
* Except for the lesions to be radiotherapy, there is at least one measurable lesion
* tumor lesions are suitable for radiotherapy
* Have previously received platinum, gemcitabine or 5-FU drugs as first-line treatment, but have not used PD-1/PD-L1 monoclonal antibody treatment
* In the 7 days before enrollment, the Child Pugh score of liver function is 7 or less

Exclusion Criteria:

* Patients with other malignant tumors
* Participated in other drug clinical trials within four weeks
* Clinical diagnosis of severe biliary obstruction or digestive tract obstruction in the past month
* Unstable angina pectoris
* Immunodeficiency
* Infectious pneumonia, non-infectious pneumonia, interstitial pneumonia
* Patients who need to use corticosteroids
* Serious chronic autoimmune diseases
* Ulcerative enteritis, Crohn's disease and other inflammatory bowel diseases
* Inflammatory and chronic diarrheal diseases such as irritable bowel syndrome;
* Sarcoidosis or tuberculosis
* Patients with hypersensitivity to human or murine monoclonal antibodies
* Pregnant and lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed according to RECIST v1.1 | 2 years
  In this trial, the International Standard (Version 1.1) developed by the entity Tumor Equipment Assessment Standard (Recist) will be used to assess objective response rate (ORR) .

SECONDARY OUTCOMES:
Progression-Free Survival, PFS | 2 years
  Reserachers use RECIST v1.1，iRECIST to assess Progression-free survival,PFS
6-month OS | 6 months
  Start calculation from the first use of drugs, researchers statistics for 6-month overal survial.
Tumor size | 2 years
  Use CT or MRI to assess the changes in tumor size

CONTACTS AND LOCATIONS:
Overall Officials: Changxian Li, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The patient's personal information involves the patient's privacy, so we do not intend to publish the patient's participant data

REFERENCES:
- [Background] Saeed A, Park R, Al-Jumayli M, Al-Rajabi R, Sun W. Biologics, Immunotherapy, and Future Directions in the Treatment of Advanced Cholangiocarcinoma. Clin Colorectal Cancer. 2019 Jun;18(2):81-90. doi: 10.1016/j.clcc.2019.02.005. Epub 2019 Feb 27. PMID 30905548
- [Background] Ilyas SI, Khan SA, Hallemeier CL, Kelley RK, Gores GJ. Cholangiocarcinoma - evolving concepts and therapeutic strategies. Nat Rev Clin Oncol. 2018 Feb;15(2):95-111. doi: 10.1038/nrclinonc.2017.157. Epub 2017 Oct 10. PMID 28994423
- [Background] Liu ZL, Liu X, Peng H, Peng ZW, Long JT, Tang D, Peng S, Bao Y, Kuang M. Anti-PD-1 Immunotherapy and Radiotherapy for Stage IV Intrahepatic Cholangiocarcinoma: A Case Report. Front Med (Lausanne). 2020 Aug 28;7:368. doi: 10.3389/fmed.2020.00368. eCollection 2020. PMID 32984358
- [Background] Sui M, Li Y, Wang H, Luo Y, Wan T, Wang X, Hu B, Cheng Y, Lv X, Xin X, Xu Q, Wang G, Lu S. Two cases of intrahepatic cholangiocellular carcinoma with high insertion-deletion ratios that achieved a complete response following chemotherapy combined with PD-1 blockade. J Immunother Cancer. 2019 May 7;7(1):125. doi: 10.1186/s40425-019-0596-y. PMID 31064408